CLINICAL TRIAL: NCT03592043
Title: A Retrospective Multicenter Canadian Registry of Patients With Mitral Regurgitation Undergoing Percutaneous Mitral Valve Repair With MitraClip
Brief Title: A Pan-Canadian, Retrospective Evaluation of MitraClip Safety and Efficacy
Acronym: PREMISE
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PREMISE
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Mitral Regurgitation
Keywords: MitraClip; Degenerative Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MitraClip: All patients who have undergone percutaneous mitral valve repair with the MitraClip system in Canada
  Interventions: Device: MitraClip

INTERVENTIONS:
Device: MitraClip — Transcatheter Mitral Valve Repair with MitraClip
  Other Names: MitraClip Clip Delivery System

SUMMARY:
The PREMISE Registry is a retrospective, observational study that will evaluate the efficacy and safety of the MitraClip in real-world Canadian practice. It will include all patients who have undergone MitraClip implantation in Canada to date.

DETAILED DESCRIPTION:
In addition to evaluating efficacy and safety, PREMISE will include a description of patient demographics, etiology of mitral regurgitation, co-morbidities, medication use and functional class. It will also compare re-hospitalization for heart failure 12 months prior and 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient has undergone percutaneous mitral valve repair with MitraClip Clip Delivery System in Canada

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have undergone percutaneous mitral valve repair with the MitraClip Clip Delivery System in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 1191 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Mitral Regurgitation (MR) severity | 12 months

SECONDARY OUTCOMES:
Hospitalization for Heart Failure | 12 months
All-cause mortality | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shamir Mehta, MD MSc FRCPC, Principal Investigator — Population Health Research Institute; McMaster University; Neil Fam, MD MSc FRCPC, Principal Investigator — St. Michael's Hospital, University of Toronto
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided